CLINICAL TRIAL: NCT05899075
Title: Evaluation of Xylitol Wipes as an Oral Hygiene Protocol for Haemophilic Children: A Randomized Clinical Trial
Brief Title: Evaluation of Xylitol Wipes as an Oral Hygiene Protocol for Haemophilic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdelmageed Mohamed Nazmy Bassiouny Mohamed Harras, BDS, Dentist at the Egyptian Ministry of Health, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 687/3906
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental)
  Interventions: Other: xylitol wipes
- group B (Placebo Comparator)
  Interventions: Other: placebo wipes

INTERVENTIONS:
Other: xylitol wipes — group A will receive xylitol wipes and group B will receive placebo wipes
  Arms: group A
Other: placebo wipes — group A will receive xylitol wipes and group B will receive placebo wipes
  Arms: group B

SUMMARY:
The purpose of this study is to evaluate xylitol wipes as an oral hygiene protocol for haemophilic children

ELIGIBILITY:
Inclusion Criteria:

* Hemophilic children A or B with No other systemic diseases.
* Aged (6-12 years).
* Co-operative.

Exclusion Criteria:

* Children on long-term antibiotics

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
dental plaque | One week
  Measure for estimating status of oral hygiene by measuring dental plaque that occurs in areas adjacent to gingival margin.

SECONDARY OUTCOMES:
Salivary levels of mutans Streptococcus | One week

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Badreldin, Study Director — AlAzhar U
Locations (1):
- AlAzhar U, Cairo, Egypt